CLINICAL TRIAL: NCT00602940
Title: The Influence of Acupuncture on Ovulation and Reproductive Hormones
Brief Title: Acupuncture for Polycystic Ovarian Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Lisa M. Pastore, UVA
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12045; NIH R21 AT002520
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2010-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; ovulation; hormones; women
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Active acupuncture treatment
  Interventions: Procedure: Acupuncture
- 2 (Sham Comparator): Sham acupuncture treatment
  Interventions: Procedure: Sham Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — 12 treatments over 8 weeks
  Arms: 1
Procedure: Sham Acupuncture — 12 treatments over 8 weeks
  Arms: 2

SUMMARY:
This is a randomized control trial of acupuncture for women with polycystic ovary syndrome. The study is triple-blinded.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-43
* confirmation of PCOS through the study
* signed informed consent
* able to receive study treatment at Virginia study sites
* agree not to use hormonal medications for the 5 months of the study

Exclusion Criteria:

* pregnant
* use of hormonal drugs 30/60 days before the study entry
* acupuncture for ovulatory disorders 30 days prior to study entry

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
ovulation in 2 out of 5 months of study participation | monthly

SECONDARY OUTCOMES:
changes in follicle stimulating hormone and luteinizing hormone | baseline vs. 2 months vs. 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Pastore, PhD, Principal Investigator — UVA OB/GYN Department
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Pastore LM, Patrie JT, Morris WL, Dalal P, Bray MJ. Depression symptoms and body dissatisfaction association among polycystic ovary syndrome women. J Psychosom Res. 2011 Oct;71(4):270-6. doi: 10.1016/j.jpsychores.2011.02.005. Epub 2011 Mar 23. PMID 21911106